CLINICAL TRIAL: NCT00657774
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled, Parallel Group, 6-Week Study to Evaluate the Effect of Multiple Doses of FlutiForm™ 250/10 Microgram HFA pMDI Twice Daily, FlutiForm™ 100/10 Microgram HFA pMDI Twice Daily, Prednisone and Placebo on the Hypothalmic-Pituitary-Adrenal Axis in Adult Subjects With Mild to Moderate Asthma.
Brief Title: A Phase I Study in Asthma Patients Evaluating the Effect of Doses of FlutiForm™ on the Amount, if Any, of Cortisol Produced by the Adrenal Glands
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SkyePharma AG (Industry)
Collaborators: Abbott (Industry)
Responsible Party: SKYEPHARMA AG, SKYEPHARMA AG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SKY2028-1-003
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2008-12-01 (Estimated); Status verified 2008-11

CONDITIONS: Asthma
Keywords: Asthma; Mild to Moderate
MeSH Terms: conditions — Asthma | interventions — fluticasone-formoterol; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): FlutiForm 250/10 ug
  Interventions: Drug: FlutiForm 250/10 ug
- 2 (Experimental): FlutiForm 100/10 ug
  Interventions: Drug: FlutiForm 100/10 ug
- 3 (Active Comparator): Oral Prednisone 10 mg
  Interventions: Drug: Oral Prednisone 10mg
- 4 (Placebo Comparator): Placebo inhaler and/or placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FlutiForm 250/10 ug — SKP FlutiForm 250/10ug is a HFA pMDI that delivers 125ug of Fluticasone propionate per actuation and 5ug of Formoterol fumarate per actuation. Patients will take 2 actuations BID for 6 weeks.
  Arms: 1
Drug: FlutiForm 100/10 ug — SKP FlutiForm 100/10ug is a HFA pMDI that delivers 50ug of Fluticasone propionate per actuation and 5ug of Formoterol fumarate per actuation. Patients will take 2 actuations BID for 6 weeks.
  Arms: 2
Drug: Oral Prednisone 10mg — 2 x 5 mg oral prednisone tablets, over encapsulated, once a day for one week.
  Arms: 3
Drug: Placebo — 2 x 5 mg placebo tablets, over encapsulated, once a day for six weeks. SKP FlutiForm placebo HFA pMDI. Two actuations BID for six weeks.
  Arms: 4

SUMMARY:
The medications being used in this study are individually approved by the Food and Drug Administration (FDA). The medication under investigation is a combination of the two medications in one inhaler. The purpose of the study is to determine how the medication affects the amount, if any, of cortisol produced by the adrenal glands.

DETAILED DESCRIPTION:
This is a Phase-1 randomized, double-blind, placebo- and active-controlled, parallel group 6 week study to evaluate the effect on the HPA axis of treatment with SKP FlutiForm 250/10 mg HFA pMDI twice daily administered over 6 weeks, FlutiForm 100/10 mg HFA pMDI twice daily administered over 6 weeks and 10 mg prednisone administered over 7 days compared to placebo. All subjects will undergo a Screening Visit to determine eligibility for the study and training on pMDI use. Eligible subjects will meet all of the following criteria: at least 6 month history of asthma, demonstrate an FEV1 of at least ≥ 60 % of predicted normal values at both Screening and Baseline visits, and stable asthma without the use of inhaled steroids for the past month or oral or parenteral corticosteroids for the past three months. All subjects will be admitted to the study site on the morning of Study Day -1 to begin a 24-hour urine collection and undergo Baseline trough PK sampling. On the morning of Study Day 1, subjects will be randomized to one of four treatment groups: SKP FlutiForm 250/10 mg twice daily + placebo capsule for six weeks, SKP FlutiForm 100/10 mg twice daily + placebo capsule for six weeks, Placebo inhaler + placebo capsule for six weeks or Placebo inhaler for six weeks + placebo capsule for 5 weeks followed by one week of 10 mg prednisone QD. After the first dose, subjects will be discharged from the study site to continue dosing at home for 6 weeks. Subjects will be required to record their compliance with their twice daily inhaler dosing and once daily oral medication dosing in a diary. Subjects will also record their predose morning and evening Peak Expiratory Flow Rate (PEFR) in a diary. Clinic visits will occur at Study Days 7, 14 and 35 during which safety assessments (AEs and vital signs) will be made, trough PK samples will be obtained and pMDI training will be continued. Also, subjects will return to the study site in the morning on Study Days 40 to 41 for observed dosing of prednisone or placebo. Subjects will be readmitted to the study site in the morning on Study Day 42 for trough PK sampling, observed dosing of prednisone or placebo and to begin a 24-hour urine collection. A safety follow-up phone call will occur 7 days later.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 at the Screening Visit;
* History of asthma for at least 6 months prior to Screening Visit
* Well controlled asthma with rescue short acting beta agonist (albuterol) and or stable doses of other medications for at least 4 weeks prior to Screening Visit
* Female subjects that are not pregnant or lactating
* Otherwise healthy as determined by the Investigator.

Exclusion Criteria:

* Life-threatening asthma within the past year or visit to emergency room for asthma in the past 3 months prior to the Screening Visit;
* Significant,nonreversible pulmonary disease (e.g. chronic obstructive pulmonary disease, cystic fibrosis or bronchiectasis)
* Use of any steroid medications, topical or inhaled steroids within 4 weeks or systemic (oral or injectable) steroids within 3 months of dosing
* An upper or lower respiratory tract infection within the last 4 weeks pior to Screening Visit or acute illness or infection within 6 weeks prior to dosing
* Any significant disease or major disorder that may jeopardize subject safety
* History of tabacco use within 6 months prior to dosing and/or smoking history > 10 pack-years
* Female subjects on hormone replacement therapy or using birth control involving hormones in the past 6 months
* Additional inclusion and exclusion criteria will evaluated by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Investigate effect of SKP FlutiForm 250/10 ug HFA pMDI BID for 6 weeks, FlutiForm 100/10 ug HFA pMDI BID, 10 mg prednisone for 7 days, compared to Placebo on the hypothalamic-pituitary-adrenal (HPA) axis using measurement of 24-hours UFC | Baseline and Study days 42-43

SECONDARY OUTCOMES:
To assess the safety profile of SKP FlutiForm HFA pMDI using incidence of adverse events (AEs) and changes in electrocardiograms (ECGs), vital signs and clinical laboratory tests. | From Baseline up to 2 weeks after last dosing

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Investigational site, Phoenix, Arizona
  - Investigational site, Anaheim, California
  - Investigational site, Long Beach, California
  - Investigational site, San Diego, California
  - Investigational site, Centennial, Colorado
  - Investigational site, Colorado Springs, Colorado
  - Investigational site, Denver, Colorado
  - Investigational site, Lakewood, Colorado
  - Investigational site, DeLand, Florida
  - Investigational Site, Pasadena, Maryland
  - Investigational site, North Dartmouth, Massachusetts
  - Investigational site, Omaha, Nebraska
  - Investigational site, Skillman, New Jersey
  - Investigational Site, Lake Oswego, Oregon
  - Investigational site, Portland, Oregon
  - Investigational site, Spartanburg, South Carolina
  - Investigational site, El Paso, Texas
  - Investigational site, New Braunfels, Texas
  - Investigational site, San Antonio, Texas